CLINICAL TRIAL: NCT01936259
Title: A Study of the Comprehensive Shoulder System With Nano Humeral Component in Total Shoulder Arthroplasty
Brief Title: Comprehensive Shoulder System Nano IDE
Acronym: Nano
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORTHO.CA.GE1.12; G110207 (Other: FDA)
Record Dates: First submitted 2013-08-23; First posted 2013-09-06 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Joint Disease
Keywords: Shoulder; Joint; Osteoarthritis
MeSH Terms: conditions — Joint Diseases; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (2):
- Comprehensive Mini Humeral Stem (Active Comparator): The Comprehensive® Shoulder System with mini stem component, which will be the control device for this clinical investigation and was 510(k) cleared under K060692 on May 30, 2006.
  The humeral stem component is manufactured from Ti6Al4V alloy. The taper has a machine finish and accepts the taper adaptor of the humeral head component. The proximal region of the bone-contacting outer surface features a porous coating of plasma-sprayed titanium alloy, while the distal portion is polished. Seventeen stem diameters are available - 4 mm to 20 mm, in 1-mm increments.
  Interventions: Device: Mini Stem
- Comprehensive Nano Humeral Component (Experimental): The stemless humeral component is manufactured from Ti6Al4V alloy. It consists of a central tapered region and six outer wings. The taper has a machine finish and accepts the taper adaptor of the humeral head component. A small groove is included just below the taper to accept an inserter/impactor. The bone-contacting outer surface features a porous coating of plasma-sprayed titanium alloy for cementless fixation in the proximal humerus. Six sizes are available - 30 mm, 32 mm, 34 mm, 36 mm, 38 mm, and 40 mm.
  Interventions: Device: Nano

INTERVENTIONS:
Device: Mini Stem — The humeral stem component is manufactured from Ti6Al4V alloy. The taper has a machine finish and accepts the taper adaptor of the humeral head component. The proximal region of the bone-contacting outer surface features a porous coating of plasma-sprayed titanium alloy, while the distal portion is polished. Seventeen stem diameters are available - 4 mm to 20 mm, in 1-mm increments.
  Arms: Comprehensive Mini Humeral Stem
Device: Nano — The stemless humeral component is manufactured from Ti6Al4V alloy. It consists of a central tapered region and six outer wings. The taper has a machine finish and accepts the taper adaptor of the humeral head component. A small groove is included just below the taper to accept an inserter/impactor. The bone-contacting outer surface features a porous coating of plasma-sprayed titanium alloy for cementless fixation in the proximal humerus. Six sizes are available - 30 mm, 32 mm, 34 mm, 36 mm, 38 mm, and 40 mm.
  Arms: Comprehensive Nano Humeral Component

SUMMARY:
The purpose of this clinical study is to determine the safety and efficacy of the Comprehensive® Shoulder System with Nano Humeral Component in Total Shoulder Arthroplasty (TSA).

DETAILED DESCRIPTION:
The purpose of this clinical investigation is to establish the safety and efficacy of the Comprehensive® Shoulder System with Nano Humeral Component in Total Shoulder Arthroplasty. Safety and efficacy of the device will be measured by collection and analysis of the following data at the two-year or greater time point (22 months post-operative or longer):

1. American Shoulder and Elbow Surgeons (ASES) Score
2. Single Assessment Numeric Evaluation (SANE)
3. Constant Score
4. Radiographic assessment of osteolysis, radiolucencies, migration, and subsidence
5. Comparison of overall adverse event rates including rates of removal/revision and other serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom the surgeon has confirmed intraoperatively, has no cyst > 1cm and not more than one cyst at the implantation site
* Patients with non-inflammatory degenerative joint disease including osteoarthritis.
* Patients where the device will be used in the correction of a functional deformity (deformities preventing congruent articulation of the glenohumeral joint)
* Patients with pain and/or loss of function in the shoulder for whom other treatment modalities have been unsuccessful.
* Patients requiring unilateral or staged bilateral shoulder arthroplasty
* Patient must be anatomically and structurally suited to receive the implants (humeral neck must be of sufficient diameter to implant at least the smallest nano humeral component and the humeral neck is intact).
* Patients who are 21-90 years of age at the time of surgery and have reached skeletal maturity.
* Patients with an ASES score ≤ 40.

Exclusion Criteria:

* Patients diagnosed with avascular necrosis or post-traumatic arthritis of the humeral head
* Patients found at the time of intraoperative examination to have a single cyst >1 cm in size or multiple cysts at the implantation site
* Patient presents with shoulder joint infection, sepsis, osteomyelitis or distant foci of infections which may spread to the implant site.
* Patients with cuff tear arthropathy.
* Patients who have undergone a Hemi-, Total, or Reverse Total Shoulder arthroplasty in the affected shoulder.
* Patient presents with a malunion or non-union of the tuberosities of the proximal humerus.
* Patients with osteoporosis, osteomalacia, rheumatoid arthritis, metabolic disorders of bone, muscle or connective tissue, gross deformity or any other condition of the proximal humerus (defined as severe destruction or deformity of the proximal humerus that precludes placement of the device) that in the Investigator's medical judgment could compromise implant fixation or bone healing.
* Rapid bone destruction, marked bone loss or bone resorption apparent on roentgenogram.
* Patients with neurologic or other disorders that would either affect the stability of the shoulder prosthesis, i.e., Charcot's joint, uncontrolled seizures, etc., or would affect their capability or willingness to return to the clinic for assessments and/or follow directions.
* Bone cancer, either primary or secondary, that affects the shoulder.
* Patients presenting with symptoms of chronic steroid use. (oral steroids for a chronic condition for 12 months prior to and including the date of surgery)
* Patients with a life expectancy of less than three years.
* Patients diagnosed with severe shoulder instability
* Patients diagnosed with subscapularis incompetence
* Patients diagnosed with any condition that may limit their ability to complete the consent form or would affect their capability or willingness to return to the clinic for assessments and/or follow directions (i.e. mental illness)
* Patients with known metal allergy
* Patients who refuse to sign the Institutional Review Board (IRB) approved consent form
* Patients who are found intraoperatively to require a specific treatment and are unable to be randomized.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2019-09-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Arizona Institute for Sports, Knees, and Shoulders, Scottsdale, Arizona
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Ortho NorthEast, Fort Wayne, Indiana
  - Orthopedic Clinic, Shreveport, Louisiana
  - Towson Orthopaedic Associates, Towson, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Buffalo, Buffalo, New York
  - Joint Implant Surgeons, New Albany, Ohio
  - Campbell Clinic Orthopaedics, Germantown, Tennessee
  - University of Virginia, Charlottesville, Virginia
  - Bon Secours St. Francis Medical Center, Midlothian, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to competitive enrollment, one extra shoulder was randomized and enrolled into the study in the Control group as the site was not aware the study had reached full enrollment.
  258 individual subjects were enrolled in the study. 7 subjects underwent study procedures bilaterally, resulting in 265 shoulders enrolled in the study.
Pre-assignment Details: Subjects were randomized 1:1 to either the Comprehensive Shoulder System with Nano Humeral Component (Investigational) or the Comprehensive Shoulder System with Mini Humeral Stem (Control). Treatment assignments occurred intraoperatively and subjects remained blinded until completion of two-year follow-up for all subjects.
Units Other Than Participants: Shoulders
Groups:
- Comprehensive Mini Humeral Stem: This arm will consist of all subjects implanted with the Control Device (Comprehensive Mini Humeral Stem).
- Comprehensive Nano Humeral Component: This arm will consist of all subjects implanted with the Investigational Device (Comprehensive Nano Humeral Component).
Period: Overall Study
Arm/Group | Comprehensive Mini Humeral Stem | Comprehensive Nano Humeral Component
Started | 130; 133 Shoulders | 131; 132 Shoulders
Completed | 118; 121 Shoulders | 111; 112 Shoulders
Not Completed | 12; 12 Shoulders | 20; 20 Shoulders

BASELINE CHARACTERISTICS:
Population: 258 individual subjects were enrolled in the study. 7 subjects underwent study procedures bilaterally, resulting in 265 shoulders enrolled in the study. Of the 7 bilateral subjects, 1 received two investigational devices, 3 received two control devices, and 3 received one of each device.
Units Other Than Participants: Shoulders
Groups:
- Total: Total of all reporting groups
Arm/Group | Comprehensive Mini Humeral Stem | Comprehensive Nano Humeral Component | Total
Number analyzed (Participants) | 130 | 131 | 258
Number analyzed (Shoulders) | 133 | 132 | 265
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.1 (9.6) | 63.1 (9.0) | 62.6 (9.3)
Sex: Female, Male [Count of Units; unit: Shoulders]
  Female | 46 | 43 | 89
  Male | 87 | 89 | 176
Race/Ethnicity, Customized [Count of Units; unit: Shoulders]
  African American | 6 | 4 | 10
  Asian | 0 | 1 | 1
  Caucasian | 125 | 126 | 251
  Hispanic or Latino | 2 | 1 | 3
Region of Enrollment [Number; unit: Shoulders]
  United States | 133 | 132 | 265
Procedure on Unilateral/Bilateral Patient [Count of Units; unit: Shoulders] — Seven subjects underwent a study procedure on each shoulder, and are classified as bilateral subjects. This measure defines how many study devices were implanted in bilateral subjects and unilateral subjects.
  Shoulders
    Bilateral | 9 | 5 | 14
    Unilateral | 124 | 127 | 251

OUTCOME MEASURES:

1. Primary Outcome: American Shoulder and Elbow Surgeon's Score (ASES)
Description: The American Shoulder and Elbow Surgeon's (ASES) Score is a tool used to measure shoulder function. The ASES score is on a scale of 0 to 100, with 0 being the worst possible score and 100 the best. The score consists of two components - pain and activities of daily living.
Time Frame: 22+ Months
Population: All subjects with ASES data available at the two year visit were assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Shoulders
Arm/Group | Comprehensive Mini Humeral Stem | Comprehensive Nano Humeral Component
Number analyzed (Participants) | 118 | 111
Number analyzed (Shoulders) | 121 | 112
score on a scale | 92.20 (13.51) | 92.47 (14.94)

2. Primary Outcome: Number of Shoulders With Absence of Revision/Removal/UADE/Fracture/Dislocation
Description: This outcome measure calculates the proportion of subjects meeting a success criteria defined in the protocol as "No unanticipated device-related adverse event, and no fracture, perforation of the bone or joint dislocation, and no fracture, perforation or dissociation of the device, and no revision or removal of any component." All subject records were evaluated for each of the disqualifying factors, and all subjects that failed at least one of the endpoint measures were identified. The success rate is defined as the number of subjects at two years not meeting any of the disqualifying factors compared to the total number of cases present at two years plus all subjects considered failures without two year data.
Time Frame: 2 years
Population: The total number of cases for each group includes all subjects with two year data, plus all subjects considered failures without two year data.
Measure: Count of Units; unit: Shoulders
Units Other Than Participants: Shoulders
Arm/Group | Comprehensive Mini Humeral Stem | Comprehensive Nano Humeral Component
Number analyzed (Participants) | 120 | 115
Number analyzed (Shoulders) | 123 | 116
Shoulders
  Success Shoulders | 114 | 107
  Failure Shoulders | 9 | 9

3. Primary Outcome: Number of Shoulders With Radiographic Success
Description: This outcome measure calculates the proportion of subjects meeting a success criteria defined in the protocol as "Subsidence of the humeral component <5 mm, and migration of the humeral component <5 mm, and no progressive lucency around the humeral component >2 mm in two or more contiguous zones, and migration of the glenoid component <5 mm, and no progressive lucency >2 mm around the entire glenoid component." All subject records were evaluated by an Independent Radiographic Reviewer (IRR) at each time point for radiographic success based on these criteria.
Time Frame: 2 years
Population: All subjects at each time point were evaluated for radiographic success based on these criteria.
Measure: Count of Units; unit: Shoulders
Units Other Than Participants: Shoulders
Arm/Group | Comprehensive Mini Humeral Stem | Comprehensive Nano Humeral Component
Number analyzed (Participants) | 130 | 131
Number analyzed (Shoulders) | 133 | 132
Shoulders
  Success Shoulders | 133 | 132
  Failure Shoulders | 0 | 0

4. Secondary Outcome: American Shoulder and Elbow Surgeon's Score (ASES)
Description: as for outcome 1
Time Frame: Pre-operative, 6 Weeks, 3 Months, 1 Year, 2 Years, 3 Years, 4 Years
Population: All subjects with an ASES score collected at each specified study time period were assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Shoulders
Arm/Group | Comprehensive Mini Humeral Stem | Comprehensive Nano Humeral Component
Number analyzed (Participants) | 130 | 131
Number analyzed (Shoulders) | 133 | 132
score on a scale
  Pre-operative | 25.8 (9.6) | 25.1 (10.7)
  6 Weeks: number analyzed (Participants) | 127 | 131
  6 Weeks: number analyzed (Shoulders) | 130 | 132
  6 Weeks | 60.1 (18.3) | 61.5 (17.4)
  3 Months: number analyzed (Participants) | 129 | 129
  3 Months: number analyzed (Shoulders) | 132 | 130
  3 Months | 80.2 (16.4) | 80.5 (15.3)
  1 Year: number analyzed (Participants) | 120 | 124
  1 Year: number analyzed (Shoulders) | 123 | 125
  1 Year | 91.2 (12.8) | 92.8 (12.2)
  2 Years: number analyzed (Participants) | 118 | 111
  2 Years: number analyzed (Shoulders) | 121 | 112
  2 Years | 92.2 (13.5) | 92.5 (14.9)
  3 Years: number analyzed (Participants) | 73 | 68
  3 Years: number analyzed (Shoulders) | 73 | 69
  3 Years | 95.0 (9.8) | 90.0 (17.8)
  4 Years: number analyzed (Participants) | 24 | 29
  4 Years: number analyzed (Shoulders) | 24 | 30
  4 Years | 95.1 (6.4) | 94.3 (11.3)

5. Secondary Outcome: Single Assessment Numeric Evaluation (SANE) Score
Description: The Single Assessment Numeric Evaluation (SANE) Score is a tool used to assess the subject's perception of their affected joint. Participants are requested to rate their shoulder function on a scale of 0 to 100, with 0 as the worst option and 100 being normal shoulder function.
Time Frame: 6 Weeks, 3 Months, 1 Year, 2 Years, 3 Years, 4 Years
Population: All subjects with a SANE score collected at each specified study time period were assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Shoulders
Arm/Group | Comprehensive Mini Humeral Stem | Comprehensive Nano Humeral Component
Number analyzed (Participants) | 130 | 131
Number analyzed (Shoulders) | 133 | 132
score on a scale
  6 Weeks: number analyzed (Participants) | 127 | 130
  6 Weeks: number analyzed (Shoulders) | 130 | 131
  6 Weeks | 55.7 (24.2) | 53.7 (23.9)
  3 Months: number analyzed (Participants) | 129 | 129
  3 Months: number analyzed (Shoulders) | 132 | 130
  3 Months | 80.4 (14.9) | 80.7 (16.1)
  1 Year: number analyzed (Participants) | 120 | 124
  1 Year: number analyzed (Shoulders) | 123 | 125
  1 Year | 90.4 (12.2) | 92.2 (9.3)
  2 Years: number analyzed (Participants) | 117 | 111
  2 Years: number analyzed (Shoulders) | 120 | 112
  2 Years | 92.3 (11.9) | 92.3 (14.5)
  3 Years: number analyzed (Participants) | 73 | 66
  3 Years: number analyzed (Shoulders) | 73 | 67
  3 Years | 94.7 (6.9) | 91.5 (15.5)
  4 Years: number analyzed (Participants) | 24 | 29
  4 Years: number analyzed (Shoulders) | 24 | 30
  4 Years | 93.4 (7.0) | 93.0 (12.9)

6. Secondary Outcome: Constant Score Adjusted for Age and Gender
Description: The Constant-Murley Shoulder Score is a scoring method used by clinicians to assess function of the shoulder. The standard score is on a scale of 0 to 100, with 0 being no shoulder function and 100 being excellent function. The age- and gender-adjusted Constant score normalizes the raw Constant score based on the subject's age and gender. The worst score on the adjusted scale is still 0, but the greatest scores can exceed 100 based on the calculations used for normalization. The scale used in this study was described by Katolik et al.
Time Frame: Pre-operative, 3 Months, 1 Year, 2 Years, 3 Years, 4 Years
Population: All subjects with a Constant score collected at each specified study time period were assessed. The score was not collected at 6 weeks to protect the subscapularis repair.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Shoulders
Arm/Group | Comprehensive Mini Humeral Stem | Comprehensive Nano Humeral Component
Number analyzed (Participants) | 130 | 131
Number analyzed (Shoulders) | 133 | 132
score on a scale
  Pre-operative | 47.2 (17.1) | 46.3 (17.1)
  3 Months: number analyzed (Participants) | 127 | 129
  3 Months: number analyzed (Shoulders) | 130 | 130
  3 Months | 82.6 (18.8) | 83.1 (19.1)
  1 Year: number analyzed (Participants) | 118 | 123
  1 Year: number analyzed (Shoulders) | 121 | 124
  1 Year | 97.9 (16.8) | 99.8 (14.9)
  2 Years: number analyzed (Participants) | 115 | 109
  2 Years: number analyzed (Shoulders) | 118 | 110
  2 Years | 100.2 (15.0) | 101.5 (16.7)
  3 Years: number analyzed (Participants) | 72 | 65
  3 Years: number analyzed (Shoulders) | 72 | 66
  3 Years | 100.2 (14.4) | 99.2 (17.3)
  4 Years: number analyzed (Participants) | 22 | 28
  4 Years: number analyzed (Shoulders) | 22 | 28
  4 Years | 98.0 (12.0) | 103.5 (15.6)

7. Secondary Outcome: Number of Shoulders Passing Radiographic Assessment of Radiolucencies and Subsidence
Description: All radiographs collected at all follow-up time points were analyzed by the Independent Radiographic reviewer. Subjects were assessed for the presence of radiolucencies considered to be failures of the radiographic co-primary endpoint (No progressive lucency around the humeral component >2 mm in two or more contiguous zones OR no progressive lucency >2 mm around the entire glenoid component) and for the presence of component subsidence. Subjects with the absence of failing radiolucencies and subsidence were considered successes.
Time Frame: 2+ years
Population: All subject radiographs at all time points that were submitted to the Independent Radiographic Reviewer were analyzed.
Measure: Count of Units; unit: Shoulders
Units Other Than Participants: Shoulders
Arm/Group | Comprehensive Mini Humeral Stem | Comprehensive Nano Humeral Component
Number analyzed (Participants) | 130 | 131
Number analyzed (Shoulders) | 133 | 132
Shoulders
  Success Shoulders | 133 | 132
  Failure Shoulders | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events reported throughout each subject's length of participation in the study are included. Length of participation is defined as the implantation date through the earlier of the date of study closure or the date of subject withdrawal, an average of 3.50 years.
Description: Subjects are counted only once in each category, even if they experienced more than one adverse event in the specified category.
Arm/Group | Comprehensive Mini Humeral Stem | Comprehensive Nano Humeral Component
All-Cause Mortality (participants affected / at risk) | 2/130 | 3/131
Serious Adverse Events (participants affected / at risk) | 55/130 | 41/131
Other Adverse Events (participants affected / at risk) | 118/130 | 105/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Comprehensive Mini Humeral Stem (N=130) | Comprehensive Nano Humeral Component (N=131)
Cardiac Arrhythmia (Cardiac disorders) | 1 (1) | 1 (2)
Death (Non-Shoulder Related) (General disorders) | 2 (2) | 3 (3)
Infection (Infections and infestations) | 2 (2) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 2 (2) | 0 (0)
Pulmonary Embolism (Vascular disorders) | 2 (2) | 0 (0)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Stroke (Vascular disorders) | 1 (1) | 1 (1)
Other General (Non-Shoulder Related) Complication (General disorders) | 44 (62) | 35 (49)
Dislocation / Subluxation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Implant or Part Failure or Fracture (Surgical and medical procedures) | 1 (1) | 0 (0)
Other Shoulder-Related Complication (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Comprehensive Mini Humeral Stem (N=130) | Comprehensive Nano Humeral Component (N=131)
Cardiac Arrhythmia (Cardiac disorders) | 2 (3) | 2 (3)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 1 (2)
Nerve Injury (Nervous system disorders) | 2 (2) | 3 (3)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (2) | 0 (0)
Other General (Non-Shoulder Related) Complication (General disorders) | 88 (193) | 72 (130)
Delayed Wound Healing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dislocation / Subluxation (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Hematoma (Skin and subcutaneous tissue disorders) | 5 (5) | 8 (8)
Humeral Fracture or Perforation (Surgical and medical procedures) | 1 (1) | 0 (0)
Implant or Part Failure or Fracture (Surgical and medical procedures) | 1 (1) | 0 (0)
Inadequate Range of Motion (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
Instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Loosening or Migration of Implants or Parts (Surgical and medical procedures) | 1 (1) | 0 (0)
Nerve Deficit (Nervous system disorders) | 0 (0) | 1 (1)
Unusual Shoulder Pain (Musculoskeletal and connective tissue disorders) | 29 (35) | 18 (23)
Wound Problems: Dehiscence, Necrosis, Drainage, Superficial Infection (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Other Shoulder-Related Complication (Musculoskeletal and connective tissue disorders) | 58 (95) | 52 (88)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator must provide the Sponsor with at least 30 days to review publications for legal and regulatory compliance and will include in publications a statement that the study was supported by the Sponsor. Sponsor confidential information will not be submitted for publication without Sponsor consent. Sponsor may request delay of publication for 60 days to allow for patent application filing.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT01936259/Prot_SAP_000.pdf